CLINICAL TRIAL: NCT05215600
Title: Anaverse™ Glenoid System and Its Instrumentation - Retrospective and Prospective, Non-Controlled Post Market Clinical Follow-Up Study
Brief Title: Anaverse™ Glenoid System and Its Instrumentation
Status: Terminated | Type: Observational
Why Stopped: Termination of PMCF study due to product discontinuation.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2017-11E
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Injuries; Shoulder Pain; Arthropathy; Arthroplasty Complications
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anaverse Shoulder System subjects: Subjects implanted with the Anaverse Shoulder System in the reversed configuration and subjects who underwent total shoulder arthroplasty conversion from anatomical to reversed.
  Interventions: Device: Anaverse Shoulder System

INTERVENTIONS:
Device: Anaverse Shoulder System — Reverse Shoulder Arthroplasty

SUMMARY:
The objectives of this study are to confirm safety, performance and clinical benefits of the Anaverse™ Glenoid System and its instrumentation by analysis of standard scoring systems, radiographs and adverse event records.

DETAILED DESCRIPTION:
The safety of the system will be assessed by monitoring the frequency and incidence of adverse events.

The performance and clinical benefits will be evaluated by assessment of the overall pain and functional performance, survival, and radiographic parameters of all enrolled study subjects.

The primary endpoint is defined by the survival of the implant system at 2 years which is based on removal or intended removal of the Anaverse™ Glenoid System baseplate and will be determined by using the Kaplan Meier method.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-75 years of age, inclusive.
* Patient is skeletally mature.
* Patient is capable of understanding the doctor's explanations, following his instructions and is able to participate in the follow-up program.
* Patient must have signed EC-approved informed consent.
* Patient requires a primary reversed total shoulder arthroplasty or a conversion from anatomical to reversed to relieve pain and restore the joint function.
* Patient has adequate quality and quantity of bone stock to support the prosthesis.
* Patient meets at least one of the following indications:

  * Advanced wear and tear of the shoulder joint resulting from degenerative, posttraumatic or rheumatoid arthritis
  * Conditions consequent to earlier operations
  * Omarthrosis or Osteoarthritis
  * Rheumatoid arthritis
  * Total joint reconstruction following trauma
* Patient has significant shoulder disability due to gross and irreparable rotator cuff deficiency. A functional deltoid muscle is necessary to use the device.
* Patient underwent reverse total shoulder reconstruction with the Anaverse Glenoid System before the date of site initiation.
* Patient has demographic, pre-operative evaluation, operative report and device information available.

Specific inclusion criteria for Conversion from Anatomical to Reversed Configuration:

* Surgery was performed with the Anaverse Glenoid System in a previously available anatomical configuration.
* Irreparable rotator cuff with superior migration of the humeral head, leading to a reduction in sub-acromial space.
* Superior tilt of the Anaverse Glenoid Baseplate not exceeding 15° compared to scapular axis.
* No evidence of mechanical or fixation failure of the Baseplate, TM Pegs or DPSC Screws, obtained pre- or intra-operatively, which would compromise the success of the conversion surgery.

Exclusion criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patient has any condition which would in the judgment of the Investigator place the patient at undue risk or interfere with the study.
* Patient is known to be pregnant or breastfeeding.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant).
* Patient has any physical conditions that would impair adequate implant support and/or prevent the use of an appropriately sized implant.
* Patient has any sign of infection (affecting the shoulder joint or in its proximity).
* Patient has glenoid presenting with large defects due to erosion, which would lead to insufficient bony support or malalignment of the devices.
* Patient is skeletally immature.
* Patient has any sign of neuromuscular compromise (excluding rotator cuff tear).
* Patient has vascular deficiency in the affected limb in sufficient degree to endanger the success of the intervention.
* Patient has absence of musculo-ligamentous supporting structures.
* Patient suffers from joint neuropathy or other conditions that may lead to inadequate skeletal fixation.
* Patient has significant injury to the upper brachial plexus.
* Patient has non-functional deltoid muscle.

Specific exclusion criteria for Conversion from Anatomical to Reversed Configuration:

* Unstable fixation of Baseplate after removal of PE Liner.
* Superior tilt of Baseplate exceeding 15° compared to scapular axis
* Superior malposition of the Baseplate which would prevent correct assembly of the Glenosphere.
* Evidence of mechanical or fixation failure of the Baseplate, TM Pegs or DPSC Screws, obtained pre- or intra-operatively, which would compromise the success of the conversion surgery.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients suffering from severe shoulder pain and disability indicated for implantation of the Anaverse™ Glenoid System in cases of total shoulder arthroplasty in reversed configuration. Patients who underwent total shoulder arthroplasty conversion from anatomical to reversed will be enrolled for subgroup analysis. Patients must meet all inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Recruitment was terminated prematurely due to early termination of the study due to product rationalization for commercial reasons. 20 participants (21 cases) of the 30 planned cases were included.
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | Anaverse Shoulder System Subjects
Started | 20; 21 Implants
Completed | 20; 21 Implants
Not Completed | 0; 0 Implants

BASELINE CHARACTERISTICS:
Population: Baseline Measures reported at participant level
Arm/Group | Anaverse Shoulder System Subjects
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 20
Height [Mean (Standard Deviation); unit: cm] | 168.3 (10.1)
Weight [Mean (Standard Deviation); unit: kg] | 80.7 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: Survival of Implant System (Kaplan Meier)
Description: The primary endpoint of this study is the survival of the implant (Reversed configuration) after 2 years, which is based on removal of the baseplate and will be determined using the Kaplan-Meier method.
Time Frame: 2 years post-op
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Anaverse Shoulder System Subjects
Number analyzed (Participants) | 20
Number analyzed (Implants) | 21
Implants | 20

2. Other Pre Specified Outcome: Constant Murley Shoulder Score (CM)
Description: The Constant Murley (CM) Score comprises outcome measures of freedom from pain (15 points), full range of function (20 points), active range of movement (40 points), and full strength (25 points). The total score is an aggregate of the individual outcome measures. The minimum score is 0 points (worst outcome), the maximum score possible is 100 points (best outcome).
Time Frame: Pre-operative (baseline), 1 year, 2 years post-operative
Population: * preoperative and 1-year data was collected retrospectively, therefore number number analyzed in the rows might differ from overall number analyzed
  * 1 patient completed study participation prior to the 2 years follow-up due to revision surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Anaverse Shoulder System Subjects
Number analyzed (Participants) | 20
Number analyzed (Implants) | 21
score on a scale
  Preop: number analyzed (Participants) | 19
  Preop: number analyzed (Implants) | 20
  Preop | 26.5 (13.5)
  1 year: number analyzed (Participants) | 7
  1 year: number analyzed (Implants) | 7
  1 year | 65.4 (17.0)
  2 years: number analyzed (Participants) | 19
  2 years: number analyzed (Implants) | 20
  2 years | 71.0 (8.9)
Statistical Analysis 1: Comparison: Anaverse Shoulder System Subjects; Test type: Other — P-values account for preoperative versus postoperative mean values at 1 and 2 years; p < 0.001, t-test, 2 sided; T-Test (Pooled)

3. Other Pre Specified Outcome: Subjective Shoulder Value (SSV)
Description: The Subjective Shoulder Value (SSV) is a single point, subjective estimate of a patient's condition. The patient is asked to rate the functionality of their operated shoulder on a scale of 0% - 100% of normal.
Time Frame: Pre-operative (baseline), 1 year, 2 years post-operative
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of normal
Units Other Than Participants: Implants
Arm/Group | Anaverse Shoulder System Subjects
Number analyzed (Participants) | 20
Number analyzed (Implants) | 21
percentage of normal
  Preop: number analyzed (Participants) | 14
  Preop: number analyzed (Implants) | 15
  Preop | 28.3 (17.5)
  1 year: number analyzed (Participants) | 9
  1 year: number analyzed (Implants) | 10
  1 year | 85.5 (11.9)
  2 years: number analyzed (Participants) | 19
  2 years: number analyzed (Implants) | 20
  2 years | 85.7 (14.0)
Statistical Analysis 1: Comparison: Anaverse Shoulder System Subjects; Test type: Other — P-values account for preoperative versus postoperative mean values at 1 and 2 years; p < 0.001, t-test, 2 sided; T-Test (Pooled)

4. Other Pre Specified Outcome: Radiographic Parameters
Description: Radiographic parameters: X-rays have been evaluated for radiolucency, osteolysis, atrophy, hypertrophy, osteophytes (glenoid), component migration (humeral implant subsidence / glenoid component migration), heterotopic ossification and scapular notching
Time Frame: Immediate post-op to 2 years post-operative
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Anaverse Shoulder System Subjects
Number analyzed (Participants) | 20
Number analyzed (Implants) | 21
Implants
  Radiolucency - Humerus ≥ 2mm: Yes | 1
  Radiolucency - Humerus ≥ 2mm: No | 20
  Radiolucency - Glenoid: Yes | 0
  Radiolucency - Glenoid: No | 21
  Osteolysis - Humerus ≥ 2mm: Yes | 1
  Osteolysis - Humerus ≥ 2mm: No | 20
  Osteolysis - Glenoid: Yes | 0
  Osteolysis - Glenoid: No | 21
  Atrophy: Yes | 0
  Atrophy: No | 21
  Hypertrophy: Yes | 0
  Hypertrophy: No | 21
  Osteophytes (Glenoid): Yes | 6
  Osteophytes (Glenoid): No | 15
  Component Migration (humeral implant subsidence / glenoid component migration): Yes | 0
  Component Migration (humeral implant subsidence / glenoid component migration): No | 21
  Heterotopic Ossification - Grade 1: Yes | 4
  Heterotopic Ossification - Grade 1: No | 17
  Heterotopic Ossification - Grade 2: Yes | 1
  Heterotopic Ossification - Grade 2: No | 20
  Heterotopic Ossification - Grade 3-4: Yes | 0
  Heterotopic Ossification - Grade 3-4: No | 21
  Scapular Notching - Grade 1: Yes | 7
  Scapular Notching - Grade 1: No | 14
  Scapular Notching - Grade 2-4: Yes | 0
  Scapular Notching - Grade 2-4: No | 21

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of surgery until study completion (up to 2 years)
Arm/Group | Anaverse Shoulder System Subjects
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaverse Shoulder System Subjects (N=20)
Infection >6 weeks (Infections and infestations) | 1 (1) — Revision surgery due to infection. Symptoms started 359 days after implantation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anaverse Shoulder System Subjects (N=20)
Urinary disorder (Renal and urinary disorders) | 1 (1)
Intraoperative humeral bone fissure (Musculoskeletal and connective tissue disorders) | 1 (1)
Traumatic Injury (Not study shoulder) (Musculoskeletal and connective tissue disorders) | 2 (2)
Instability - Luxation (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this study are the low sample size of 21 cases as well as the short follow-up period of two years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT05215600/Prot_SAP_001.pdf